CLINICAL TRIAL: NCT01403441
Title: Radiosurgical Neuromodulation for Refractory Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Potential AE
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Hugh Brent Solvason, Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-12012010-7249; eprotocol 10186
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Bipolar Disorder
Keywords: Refractory Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Precision radiotherapy is delivered on Day 1 using the Cyberknife System to Brodmann area cingulate 25.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiosurgical Neuromodulation (Experimental): Bilateral Radiosurgical Neuromodulation using the Cyberknife
  Interventions: Device: Radiosurgical Neuromodulation using the Cyberknife

INTERVENTIONS:
Device: Radiosurgical Neuromodulation using the Cyberknife — our team has selected 60 Gray (Gy) as the dose to the target margin to be used for radiosurgical neuromodulation in patients with intractable bipolar disorder; the target being the anterior cingulate (Cg) that correlates with Brodmann area 25 (Cg25).

SUMMARY:
This study is designed to evaluate the safety and effectiveness of an investigational procedure for treating people with treatment resistant bipolar depression (TRD). Precise dose delivery of radiation to the predetermined targets in the brain will be accomplished with known Cyberknife stereotactic radiosurgery methods. This technology is considered to be noninvasive (does not physically invade your body). We will be studying if the Cyberknife influences the sensitivity of certain nerves of your brain. Although many clinical treatments for psychiatric conditions have been done using stereotactic radiosurgery, the present study is experimental, because we are seeking to use more moderate doses of radiation that are intended not to destroy any brain cells, but to normalize or modulate their function.

DETAILED DESCRIPTION:
Main objective: To determine the safety of Radiosurgical Neuromodulation (RSN) for Refractory Depression using X-rays in a population of subjects with severe treatment resistant bipolar depression over a 12-month observational period post treatment. While almost any radiosurgical device could be used, the research team has extensive experience with the Accuray CyberKnife System, K011024, and it will be used for planning and delivery of the 6 megavolt (MV) X-ray treatment for this study.

Participation will be dependent upon subjects having a diagnosis of bipolar depression and meeting criteria for treatment resistance. Treatment resistance will be defined as a failure to show clinical improvement after at least four different medication trials and/or one course of electroconvulsive therapy (ECT) during the current episode. A medication trial is defined as an adequate dose and duration of one of four classes of psychoactive medications: lithium, anticonvulsant mood stabilizers, atypical antipsychotic mood stabilizers, and/or antidepressant medications. One course of ECT is defined as receiving six acute treatments. The study will include subjects who have failed ECT, or have had intolerable side effects to ECT, or elected not to receive such treatment due to stigma, or concern over possible side effects of the ECT treatment itself. The subjects enrolled will have exhausted all reasonable treatment strategies, and currently have no other reasonable or viable treatment options for their illness.

Secondary objective: To examine clinical outcome initially over 3 months, then with follow up at 6, 9 and 12 months. Depression will be assessed using the Hamilton Depression Rating Scale (HDRS) 24 item, while manic symptoms will be measured by using the Young Mania Rating Scale (YMRS), and the Clinical Global Impression of Severity of illness (CGI-S), and Improvement (CGI-I). A battery of neuropsychological tests will be administered as well, assessing memory with the California Verbal Learning Task (CVLT), prefrontal function using a Delas-Kaplan Executive Function System (DKEFS) battery including the DKEFS Sorting task, DKEFS Trails task, DKEFS color-word interference task, and the DKEFS verbal fluency task. In addition, the investigators will request information regarding any possible adverse events that occur during this trial.

The intended use for the CyberKnife System, the radiosurgical device being used in this research study, is to administer radiomodulation to the cingulate cortex target Cg25 in patients with refractory bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate, all patients must meet the following criteria:

* Men and women 22-65 years of age
* Primary diagnosis of bipolar depression, as per the Diagnostic and Statistical Manual - Text Revision (DSM IV-TR) criteria
* The current major depressive episode has been for at least one year
* Hamilton Depression Rating Scale (HDRS)-24 item greater than or equal to 20
* Negative urine pregnancy in female subjects
* No current psychotic symptoms
* No comorbid post traumatic stress disorder, the inclusion of subjects with other psychiatric comorbidity will be determined by the investigator prior to enrollment
* No personality disorder that in the opinion of the investigator may compromise the subjects ability to participate and be compliant with the elements and procedures of the study
* No substance abuse of dependence in the last 6 months
* A negative urine drug screen
* On a stable dose of their current medication regimen for four weeks
* Treatment resistance: A history of failure to show clinical improvement after at least four different medication trials of adequate duration and dose and one course of ECT. A course of ECT is not mandatory for those who have declined the procedure due to stigma, patient preference, or intolerance. One course of ECT is defined as receiving six acute treatments. (Note: the Antidepressant Treatment History Form (ATHF) does not apply to bipolar depression where mood stabilizers are the treatments of choice in the first three steps in an algorithm to treat bipolar depression)
* No available reasonable treatment options at the time of enrollment
* Competent to understand the risks and potential benefits of the study
* Able to provide written informed consent for the full screening phase, as well as the treatment period of the protocol, including the baseline MRI, CT and positron emission tomography (PET) imaging
* Signed consent form for participation in the study

Exclusion Criteria:

Patients who meet the following criteria will be excluded from participation in this research study:

* Rapid cycling bipolar illness
* History of schizophrenia, schizoaffective disorder, or psychosis
* Severe suicidal thoughts that may put the subject at risk of either an attempted suicide or completed suicide for the duration of the trial, as determined by the investigator at the time of enrollment
* Current substance abuse or in the process of withdrawal from mind-altering substances including alcohol, stimulants, or sedatives
* Undisclosed or undiagnosed unstable medical or neurologic illness including stroke, significant brain malformation, brain mass
* Previous whole-brain radiation
* Brain-implanted devices such as deep brain stimulation leads, aneurysm clips
* A history of seizure disorder
* History of moderate to severe brain injury
* Current treatment with either metronidazole or cisplatinum and an inability to discontinue prior to RSN
* Pregnancy or breast feeding
* Unstable medical illness
* Current participation in another investigational trial or participation within 30 days of enrollment

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Brent Solvason, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in August 2010, through July 2012. Subjects recruited from outpatient referrals. 5 subjects were screened, 3 enrolled.
Pre-assignment Details: No group assignment, open label study.
Groups:
- Open Treatment Study: All three subjects had Cyberknife treatment targeting the subgenual cingulate cortex, and then followed for 12 months observation and assessments of depression severity.
Period: Overall Study
Arm/Group | Open Treatment Study
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treatment Resistant Depression
Groups:
- Open Treatment Study: Open treatment with Cyberknife System targeting brain area cingulate 25.
Arm/Group | Open Treatment Study
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Event
Description: An event that required hospitalization due to an unanticipated worsening of the subjects bipolar disorder.
Time Frame: Baseline and 12 months.
Population: Patients with bipolar disorder in the depressive phase who have not responded to any available treatment
Measure: Number; unit: event
Groups:
- Radiosurgical Neuromodulation: Bilateral Radiosurgical Neuromodulation using the Cyberknife
  Radiosurgical Neuromodulation using the Cyberknife: our team has selected 60 Gy as the dose to the target margin to be used for radiosurgical neuromodulation in patients with intractable bipolar disorder; the target being the anterior cingulate that correlates with Brodmann area 25 (Cg25).
Arm/Group | Radiosurgical Neuromodulation
Number analyzed (Participants) | 3
event | 1

2. Secondary Outcome: Hamilton Depression Rating Scale (HDRS) - 17 Item
Description: The HDRS is a rating scale measures the severity of depressive symptoms. The scale consists of 17 symptoms with severity anchors that are scored from 0 to 4. The maximum score (most severe depression) is 68, the lowest (no depressive symptoms) is 0.
Time Frame: Baseline and 12 months
Population: Patients with Bipolar disorder in the depressive phase that have not responded to available treatments
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open Treatment Study: All three subjects had Cyberknife treatment, and then followed for 12 months observation and assessments.
Arm/Group | Open Treatment Study
Number analyzed (Participants) | 3
units on a scale | 24.0 (2.0)

3. Secondary Outcome: Clinical Global Impression - Severity (CGI-S) at Baseline and 12 Months
Description: The CGI-S assess the overall severity of depression over the 12 month observation period following Cyberknife System. It is rated from 1 (well or remitted) to 7 (severely ill, among the most depressed).
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open Treatment Study: Subjects had precision targeted radiotherapy using the Cyberknife System that targeted the subgenual cingulate cortex (approximating Brodmann area 25), and then had assessments of depression severity at intervals for 12 months.
Arm/Group | Open Treatment Study
Number analyzed (Participants) | 3
units on a scale
  12 month | 3 (1.2)
  Baseline | 6 (1.0)

4. Secondary Outcome: Delis-Kaplan Executive Function System (D-KEFS) Composite Score
Description: D-KEFS is a neurocognitive assessment of executive function. The composite score is derived from scores on tests that include Trails A, Color Word Interference, Verbal Fluency, Sorting, WAIS III Digit Span, and CVLT II Long Delay Free Recall. The scores are reported as deviation from a mean of 10, with a standard deviation of 3. A score of 7 is one standard deviation below the mean, while a score of 13 is 1 standard deviation above the mean. Higher numeric outcomes reflect better performance on the test, lower values reflect poorer performance. Results reflect scores at baseline, and 12 month observation period following Cyberknife System
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Treatment Study
Number analyzed (Participants) | 3
units on a scale
  Baseline | 8.4 (2.2)
  12 months | 11.8 (2.5)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Radiosurgical Neuromodulation: Precision stereotactic radiotherapy targeted the subgenual cingulate cortex (which approximates Brodmann area cingulate 25) using 60 Gy as the dose to the target margin using the CyberKnife System.
  Subject 3 had a signal abnormality on the MRI of the brain at 9 month time point which was unchanged 12 months on both T1 and T2 acquisition images. This is one adverse event that was sustained. The presence of the signal abnormality at 9 and 12 months indicates it did not change. A change in this type of signal abnormality would not be expected to resolve on that time scale. This adverse event is one occurrence that sustained for the next 3 months.
Arm/Group | Radiosurgical Neuromodulation
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiosurgical Neuromodulation (N=3)
Psychotic mania (Nervous system disorders) | 1 (1) — The patient self-discontinued Symbyax after 6 months in the study. He had remitted at this point, and felt he did no longer needed this medication, and it was too expensive. He subsequently became hypomanic then manic and required hospitalization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiosurgical Neuromodulation (N=3)
Signal Abnormality on MRI (Nervous system disorders) | 1 (1) — Subject 3 had a signal abnormality in the subgenual cingulate cortex on both T1 and T2 images at 9 and 12 months

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No